CLINICAL TRIAL: NCT00218465
Title: A Double-Blind, Placebo-Controlled Trial of the NMDA Glycine Site Antagonist, GW468816, for Prevention of Relapse to Smoking
Brief Title: Effectiveness of GW468816, an NMDA Glycine Site Antagonist, for Prevention of Relapse to Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Mclean Hospital (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Maurizio Fava, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIDA-19378-2; U01DA019378 (NIH); IND 74964 (Other: IND Number)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Nicotine Dependence
Keywords: Drugs, Investigational; Therapies for Relapse to Nicotine; Relapse Prevention; Nicotine Cessation Therapies; Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — GW 468816

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GW468816 (Experimental): Glycine Antagonist GW468816, 200 mg/day, for a 5-week trial
  Interventions: Drug: GW468816
- Placebo (Placebo Comparator): Placebo, 200 mg/day, for a 5-week trial
  Interventions: Drug: Placebo Comparator: Placebo

INTERVENTIONS:
Drug: GW468816 — Pharmacotherapies for Relapse Prevention
  Other Names: GW468816: NMDA glycine-site antagonist
  Arms: GW468816
Drug: Placebo Comparator: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of the glycine antagonist, GW468816, compared with placebo on duration of abstinence and rates of relapse in recently quit female smokers in a randomized, double-blind, five-week clinical trial.

According to the investigators, the new medication, GW468816, is thought to send certain signals in the brain that may be effective in helping people stay abstinent after they have recently quit smoking. GW468816 is a non-nicotine drug.

The investigators of this study hypothesize that subjects receiving GW468816 will demonstrate a significantly longer time to relapse to smoking than those in the placebo group, as measured by the primary outcome measure (see below).

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable mortality in developed countries. Pharmacotherapy, including bupropion and nicotine replacement therapy (NRT), is universally recommended for smoking cessation treatment; however, even with treatment, the majority of smokers either fail to quit in the short term or relapse in the first year. The high failure rate reported for smoking cessation, then, presents a challenge to explore innovative approaches to treating relapse to smoking.

The purpose of this study, then, is to evaluate the efficacy of the glycine antagonist, GW468816, compared with placebo on duration of abstinence and rates of relapse in female outpatient smokers during a randomized, double-blind, five-week clinical trial.

To do this, the investigators will conduct a two-phase study, in which 300 adult, female outpatient smokers will be enrolled.

Phase I will consist of an 8-week smoking cessation study in which nicotine replacement therapy (NRT) and a behavioral intervention are openly administered on a tapered schedule. Participants who are able to quit smoking after 7 weeks in this preliminary study will then be eligible to enter Phase II.

Phase II is a 5-week, double-blind, placebo-controlled, relapse prevention trial with the investigational medication, GW468816.

Participants in the Phase I smoking cessation study will begin by receiving nicotine replacement therapy in the form of the patch and brief support to stop smoking. Participants will be required to schedule office visits every 1-2 weeks throughout Phase I.

Subjects who are abstinent at the end of Phase I will be eligible to continue Phase II, in which they will be randomly assigned by chance to receive the investigational medication, GW468816, at 200 mg or placebo (a pill that looks exactly like the study drug but contains no active drug). Participants will be required to schedule weekly office visits throughout Phase II.

Subjects who complete the 15-week trial (both Phases I and II) will enter the 6-Month Follow-Up to evaluate rates of long term abstinence from nicotine. They will have office visits at Weeks 20, 24, 28, 32, 36, and 40 after discontinuation of study medications.

Participants who enter the study will be offered the opportunity to participate in an ancillary neuroimaging study of mechanisms and surrogate markers of relapse that includes BOLD fMRI and MR spectroscopy, to be carried out at the McLean Brain Imaging Center.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. WOMEN aged 18-65 years, inclusive
3. Self-report of smoking 10 or more cigarettes per day in the past 6 months and expired air CO >10 ppm at the time of enrollment
4. DSM-IV criteria for current Nicotine Dependence satisfied
5. Subjects must be willing to take the study medication and be motivated to quit smoking (willing to set a quit date within 2 weeks of entry into the protocol)
6. Women of childbearing potential must have a negative urine pregnancy test (quantitative HCG) at baseline and at week 8, prior to receiving the first dose of study medication and females must agree to use an approved form of contraception from the day of the first dose of study medication for 90 days after the last dose of study medication. Approved forms of contraception include any of the following:

   * Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, through the treatment phase and for 90 days after discontinuation of study medication.
   * Sterilization of male partner
   * Implant of levonorgestrel
   * Injectable progesterone
   * Intrauterine device (IUD) with <1 percent rate of failure per year
   * Any other method with published rate of failure of <1 percent per year Due to induction of cytochrome p450 3A4, oral contraceptives may be continued during the study but cannot be relied upon as a sole means of contraception, and a second method of contraception such as a barrier method will be required and reimbursed by the study.

Exclusion Criteria:

1. Pregnant or able to become pregnant and not willing to use approved contraception
2. Severe unstable medical illness including cardiovascular, hepatic, renal, respiratory, metabolic, neurological, or hematological disease by history, physical examination or clinical laboratory test results such that hospitalization for treatment of that illness is likely within the next two months
3. Life-threatening arrhythmia, cerebro-vascular or cardiovascular event within six months of enrollment
4. Elevation over 1.5 times upper limit of normal value (ULN) of any of the following laboratory results: Total, conjugated, or unconjugated bilirubin; alkaline phosphatase, alanine transferase (ALT), aspartate aminotransferase (AST), creatine phosphokinase (CPK), or lactate dehydrogenase (LDH).
5. Use of tobacco-containing products other than cigarettes (e.g., cigar, pipe)
6. Abuse or dependence of any substance other than nicotine or caffeine in the past 6 months. Abuse of alcohol is here defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than two units (females). One unit is equivalent to a half-pint (220mL) of beer or one (25mL) measure of spirits or one glass (125mL) of wine.
7. Diagnosis of major depressive disorder in the past 6 months
8. Lifetime DSM-IV diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, bipolar disorder, delusional disorder or psychotic disorders not elsewhere classified
9. History of non-response in the past month to an adequate trial of nicotine re placement therapy, defined as nicotine replacement > 21 mg per day patch (or equivalent dose of gum, inhaler, nasal spray, or lozenge) for at least 4 weeks.
10. History of multiple adverse drug reactions
11. Use of an investigational drug or device within 4 weeks of enrollment
12. Concurrently enrolled in a study that involves exposure to a drug or device.
13. Urine positive for drugs of abuse at screening visit.
14. Use of statins during the period of the investigation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, M.D., Principal Investigator — Massachusetts General Hospital; Eden Evins, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Brain Imaging Center, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- 816 Group: Glycine Antagonist GW468816, 200 mg/day, for a 5-week trial.
- Placebo: Placebo group for 5 week relapse prevention trial.
Period: Overall Study
Arm/Group | 816 Group | Placebo
Started | 50 | 48
Completed | 33 | 30
Not Completed | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 816 Group | Placebo | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 48 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (10.5) | 46.5 (10.4) | 47.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse to Smoking in the 5-week Relapse Prevention Phase.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 816 Group | Placebo
Number analyzed (Participants) | 50 | 48
days | 14.5 (14.0) | 12.4 (12.5)

2. Primary Outcome: Number of Abstinent and Nonabstinent Participants at End of 5 Week Placebo-controlled Relapse Prevention Trial
Time Frame: 5 weeks
Measure: Number; unit: participants
Arm/Group | 816 Group | Placebo
Number analyzed (Participants) | 50 | 48
participants | 50 | 48

3. Primary Outcome: Days to Relapse Within the 60 Days Following Randomization
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 816 Group | Placebo
Number analyzed (Participants) | 50 | 48
days | 20.8 (18.3) | 20.6 (20.3)

ADVERSE EVENTS:
Time Frame: Five weeks.
Arm/Group | 816 Group | Placebo
Serious Adverse Events (participants affected / at risk) | 2/50 | 1/48
Other Adverse Events (participants affected / at risk) | 31/50 | 31/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 816 Group (N=50) | Placebo (N=48)
small cell adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
facial edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 816 Group (N=50) | Placebo (N=48)
Cardiovascular (Cardiac disorders) | 3 (3) | 2 (2)
General/Administration Site (General disorders) | 8 (8) | 7 (7)
Gastrointestinal (Gastrointestinal disorders) | 14 (14) | 11 (11)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Nervous System (Nervous system disorders) | 12 (12) | 15 (15)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (13)
Dermatological (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No